CLINICAL TRIAL: NCT00396695
Title: Neuroimmunological Model of Traumatic Memory
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Other Study IDs: HP 6-198 R
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2006-11

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD, traumatic memory
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: Blood test

SUMMARY:
Traumatic events may lead to strong emotional episodic memories common in Post- Traumatic Stress Disorder(PTSD). Intense affect may inhibit efficacy of glutamatergic neurotransmission in two particular areas of the limbic system that have been implicated in the processing of emotionally charged memories: the amygdala and the hippocampus(1,2).

Dysfunction of glutamatergic neurotransmission is associated with disbalance of long-term potentiation (LTP) and long-term depression (LTD)- two underlying mechanisms that cooperate to achieve synaptic plasticity and its expressations- learning and memory(3). LTP- the long lasting enhancement of synaptic function includes changes in the amount of neurotransmitter glutamate released into a synapse, changes in the levels of key proteins in synapses, protein phosphorylation and changes the density of receptors on their synaptic membranes. LTD is the inverse of LTP, a long lasting reduction in synaptic transmission (4). Interactions among the different forms of plasticity underlie different forms of memories. Normally these mechanisms are balanced.

In the current literature there is data that a class I major histocompatibility complex (MHC class I) molecules, known to be important for immune responses to antigen, are expressed also by neurons that undergo activity-dependence, long-term structural and synaptic modifications (5). The brain produces its own immune molecules, the proteins MHC class I and CD3-zeta (a component of receptors for MHC class I). In the immune system, the two proteins act as part of a lock and key system to recognize and get rid of the body's foreign invaders. The CD3-zeta polypeptide is component of the T cell antigen receptor (TCR) which contribute to its efficient cell surface expression and account for part of its transducing capability (6).

In the brain, they may be part of a signaling system that recognizes and eliminates inappropriate neural connections. Expression of MHC class I is regulated by the naturally occurring electrical activity, and sensitive to both natural and pathological changes in the activity. Electrical activity of neurons drives to an establishment of the final pattern of connection. Changes in the strength of individual synapses such as potention and depression leads to stabilization and withdrawal, respectively, of the affected connections. There are data, that in mice with deficiency of MHC class I and CD3-zeta the LTP in the hippocampus is enhanced significantly and LTD is absent. Thus, MHC class I is crucial for translating activity into changes in synaptic strength and neuronal connectivity in vivo. He required for normal activity dependent potentiation, depression, removal of inappropriate connection and responding to injury in the CNS (6).

Glutamate receptors play critical roles in LTP/LTD mechanisms. Some researchers consider that a key role in pathogenesis of PTSD is being played by excessive excitation of NMDA-receptors in limbic system structures (1). The existing data allows to assume, that equation of plasticity mechanisms depends on mutual relations between the MHC class I and glutamate receptors.

T-cells, like neurons, express high levels of glutamate receptors that are identical to the brain glutamate receptors. Presence of ionotropic and metabotropic glutamate receptors in membranes of lymphocytes makes them sensitive to the same alarm molecules which operate neuronal activity. Glutamate by itself triggers several T-cell activation which differs quantitatively or qualitatively from that ones triggered by "classical' T-cell activators like antigens(7). There are data about influence of T cell receptor-CD3 complex- on the expression of T-cells glutamate receptors (8). It is possible, that the key roles in this function play CD3-zeta.

DETAILED DESCRIPTION:
Working hypothesis and aims

Trauma-related LTP/LTD disbalance in favor of potentaion and excessive excitation of glutamate receptors generated when arousing experiences occur in conjunction with memory-related activation of the hippocampus and amigdala. Traumatic memories connected to the amplification of mechanism LTP, when new information is unable to induce reliable LTD, which reverses synaptic plasticity formed during previous emotional learning experiences.

MHC class I and CD3-zeta play a key role in these changes. We assume that the composition of glutamate receptors and CD3-zeta expression in T-cells can be used as the model reflecting for LTP/LTD balance in CNS.

The work includes the learning of following parameters:

1. The Expression in T-cells: glutamate receptors, CD3-zeta.
2. Glutamate level in plasma
3. Cytokines levels in plasma:

   1. interferon-γ that can induce some components of class I MHC (9).
   2. tumor necrosis factor-α that influences the AMPAR expression and plays a role in LTP reduction (10).

Groups (of 20 people each) will make patients with a priori various degree of LTP/LTD balance: healthy people and PTSD patients.

People suffering PTSD, frequently have conditions when they again, brightly and deeply experience event injuring them. The memoirs painted by painful emotions, seize attention of the person and then it seems to him as if he again experiences injuring event and sees it as real.

We assume, that it is connected to the unable to induce reliable LTD, and that the composition of glutamate receptors and CD3-zeta expression in T-cells such people should differ from healthy.

Used method: enzyme- linked immunosorbent assay (ELISA), FACS

ELIGIBILITY:
Inclusion Criteria:

* male and female between 18-60 years
* PTSD

Exclusion Criteria:

* any immune system disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2006-10; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Mizruchin, MD, Principal Investigator — Sieff Government Hospital
Locations (1):
- Sieff Government Hospital, Safed, Israel

REFERENCES:
- [Background] Heresco-Levy U, Kremer I, Javitt DC, Goichman R, Reshef A, Blanaru M, Cohen T. Pilot-controlled trial of D-cycloserine for the treatment of post-traumatic stress disorder. Int J Neuropsychopharmacol. 2002 Dec;5(4):301-7. doi: 10.1017/S1461145702003061. PMID 12466030
- [Background] Bessel van der Kolk. Memory and the evolving psychobiology of post traumatic stress. 1994.
- [Background] Bellone C, Luscher C. mGluRs induce a long-term depression in the ventral tegmental area that involves a switch of the subunit composition of AMPA receptors. Eur J Neurosci. 2005 Mar;21(5):1280-8. doi: 10.1111/j.1460-9568.2005.03979.x. PMID 15813937
- [Background] Gaiarsa JL, Caillard O, Ben-Ari Y. Long-term plasticity at GABAergic and glycinergic synapses: mechanisms and functional significance. Trends Neurosci. 2002 Nov;25(11):564-70. doi: 10.1016/s0166-2236(02)02269-5. PMID 12392931
- [Background] Boulanger LM. MHC class I in activity-dependent structural and functional plasticity. Neuron Glia Biol. 2004 Aug;1(3):283-9. doi: 10.1017/S1740925X05000128. PMID 18185853
- [Background] Malissen M, Gillet A, Rocha B, Trucy J, Vivier E, Boyer C, Kontgen F, Brun N, Mazza G, Spanopoulou E, et al. T cell development in mice lacking the CD3-zeta/eta gene. EMBO J. 1993 Nov;12(11):4347-55. doi: 10.1002/j.1460-2075.1993.tb06119.x. PMID 8223444
- [Background] 7. Mia Levite. Direct Bi-Directional Dialogues Between The Nervous System And The Immune System in health and disease. www.weizmann.ac.il/neuro 2006.